CLINICAL TRIAL: NCT03176017
Title: Ejaculatory Sparing Transurethral Incision Of The Prostate (ES-TUIP) Versus Conventional TUIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HoLES-TUIP
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-09

CONDITIONS: Prostate Hyperplasia; Transurethral Incision Of The Prostate; Ejaculatory Dysfunction
Keywords: Transurethral Incision Of The Prostate; Prostate; Ejaculatory Sparing
MeSH Terms: conditions — Prostatic Hyperplasia; Ejaculatory Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ejaculatory sparing TUIP (Active Comparator): Ejaculatory sparing TUIP
  Interventions: Procedure: Ejaculatory sparing TUIP
- Conventional TUIP (Placebo Comparator): regular non ejaculatory sparing TUIP
  Interventions: Procedure: Conventional TUIP

INTERVENTIONS:
Procedure: Ejaculatory sparing TUIP — The bladder neck will be incised and vaporized at the 5 or 7-o'clock position. The incision will start near the ureteral orifice and carry downward to about 0.5-1.0 cm proximal to the verumontanum
  Other Names: ES-TUIP
  Arms: Ejaculatory sparing TUIP
Procedure: Conventional TUIP — the bladder neck will be incised by Collins knife at the 5 or 7-o'clock position till the verumontanum.
  Other Names: regular non ejaculatory sparing TUIP
  Arms: Conventional TUIP

SUMMARY:
In this study, Investigators planned to compare ejaculatory sparing and non-ejaculatory sparing (conventional) TUIP using both subjective and objective assessment tools for the degree of deobstruction.

Furthermore, the impact of both techniques on ejaculation and its secondary effect on orgasm perception and different domains of sexual function will be thoroughly assessed.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) score ≤3.
* TRUS estimated prostate weight ≤ 35 grams.
* Sexually interested and having continuous relationship with the same partner (interested).
* Bladder outlet obstruction index (BOOI ) ≥ 20 as per pressure flow study

Exclusion Criteria:

* Preoperative sexual or ejaculatory disturbances or pelvic pain syndrome
* Neurological disorders that can affect potency and ejaculation e.g. long standing uncontrolled diabetes mellitus (DM) type 2 (> 10 years), DM type 1, cerebral stroke, Parkinsonism
* Urodynamic changes consistent with urethropathy or detrusor hypocontractility
* Previous pelvic surgeries or radiotherapy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
impact on ejaculatory function and subsequently the impact of reported ejaculatory changes on orgasm perception | 1 year
  Ejaculatory domain of Male sexual health questionnaire (Ej-MSHQ)

SECONDARY OUTCOMES:
Erectile function domains (erectile function, orgasm, desire, intercourse satisfaction and overall satisfaction) | 1 year
  International index of erectile function-15 (IIEF-15) questionnaire
Patient reported functional urinary outcomes | 1 year
  International prostate symptom score (IPSS) questionnaire
maximum flow rate (Q.max) | 1 year
  milliliters per second.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shoma, MD, Study Chair — Urology and Nephrology center; Nasr Eltabey, MD, Study Director — Urology and Nephrology center; Ahmed N Elshal, MD, Study Director — Urology and Nephrology center; Mahmoud Laimon, Msc, Principal Investigator — Urology and Nephrology center; Ahmed Elkashef, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes meta-analyses by contact the Dr Ahmed Elshal, MD (Study Chair)